CLINICAL TRIAL: NCT06548412
Title: CTX-009 With Gemcitabine, Cisplatin, and Durvalumab as First-line Therapy in Patients With Unresectable or Metastatic Biliary Tract Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Compass Therapeutics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0279; NCI-2024-06735 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead-in: CTX-009+ Durvalumab+Gemcitabine+cisplatin (Experimental): Participants will be administered treatment on an outpatient basis
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Drug: CTX-009
- Expansion: CTX-009+ Durvalumab+Gemcitabine+cisplatin (Experimental): Participants will be administered treatment on an outpatient basis
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Drug: CTX-009

INTERVENTIONS:
Drug: Gemcitabine — Given by IV
Drug: Cisplatin — Given by IV
Drug: Durvalumab — Given by IV
Drug: CTX-009 — Given by IV

SUMMARY:
To evaluate combination therapy of adding CTX-009 to the standard therapy GCD as first-line therapy in patients with unresectable or mBTC.

DETAILED DESCRIPTION:
Primary Objectives:

1. Assess tolerability/safety of this combination and determine the maximum tolerated dose (MTD) of CTX-009.
2. Assess 6 month progression-free survival to the combination therapy according to RECIST 1.1

Secondary Objectives:

1. Assess objective response rate (ORR)
2. Assess duration of response (DOR)
3. Assess overall survival (OS)
4. Assess progression free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of CTX-009 in combination with durvalumab, gemcitabine, and cisplatin in patients <18 years of age, children are excluded from this study.
2. Ability to understand and the willingness to sign a written informed consent document.
3. Histologically or cytologically confirmed (outside pathology reports will be accepted) unresectable advanced, metastatic, or recurrent BTC at the time of enrollment that has not been previously treated in the metastatic setting.
4. Patients must have measurable disease per RECIST v1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
5. ECOG performance status ≤2
6. Patients must have adequate organ and marrow function within 14 days of treatment as described below (patients must be free of G-CSF treatment within 14 days prior to the lab test)

   * absolute neutrophil count ≥1,000/mcL
   * platelets ≥100,000/mcL
   * Hemoglobin ≥ 9 g/dL.
   * WBC ≥ 3,000/mm3
   * total bilirubin ≤ 1.5 institutional upper limit of normal (ULN)
   * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN (≤5×ULN w/ hepatic metastasis)
   * Calculated creatinine clearance ≥ 60mL/min (determined as per Cockcroft-Gault)
   * Urine protein ≤ 1+ by dipstick
   * Serum amylase and lipase level ≤ 1.5 X ULN
   * Serum albumin ≥ 3.0 g/dL
7. No evidence of ongoing active infection.

   * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
   * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
8. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Patients with asymptomatic and controlled brain cancer are eligible for inclusion if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
9. The effects of CTX-009 on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after completion of CTX-009 administration. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

   * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
   * History of hysterectomy or bilateral salpingo-oophorectomy.
   * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
   * History of bilateral tubal ligation or another surgical sterilization procedure.
   * Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of CTX-009 administration.

Exclusion Criteria:

1. Previous treatment of the current malignancy. Patients who received prior perioperative treatment (adjuvant and neoadjuvant) are eligible.
2. History of active interstitial lung disease.
3. History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, or evidence of active pneumonitis on baseline imaging
4. Major surgical intervention within 28 days of Day 1 (Biliary stent placement, biliary stent exchange, and Endoscopic retrograde cholangiopancreatography (ERCPs) are not considered major surgical interventions)
5. Patients with percutaneous transhepatic biliary drains (PTBD)
6. Symptomatic or uncontrolled central nervous system (CNS) metastasis (However, patients with asymptomatic CNS metastasis can participate provided that systemic corticosteroid treatment was discontinued at least 4 weeks prior to screening and that the patient is radiologically and neurologically stable or improving). Unless symptomatic, imaging of the head is not required for screening.
7. Has an active infection requiring systemic therapy, with the exception of HBV and HCV
8. Known positive serology for HIV (Human immunodeficiency virus)
9. A history of the following hemorrhage-related or gastroenterological disease:

   * Active hemorrhage, hemorrhagic diathesis, coagulopathy, or tumor in great arteries
   * History of clinically significant gastroenterological disease, such as peptic ulcer, GI bleeding, GI or non-GI fistula, perforation, abdominal abscess, clinical symptoms, and signs of GI obstruction, need for parenteral hydration or nutrition, or inflammatory bowel disease (IBD)
10. Active, uncontrolled autoimmune disease that might deteriorate when receiving an immune-stimulatory agent. Patients with vitiligo, psoriasis, primary sclerosing cholangitis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
11. Active, uncontrolled inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
12. Patients who received antiplatelet drugs (aspirin, clopidogrel, etc.) or anticoagulant drugs (warfarin, heparin, etc.) within 2 weeks prior to screening, or is expected to need those drugs during the clinical study.
13. A history of the following cardiovascular diseases in past 5 years:

    * Congestive heart failure (CHF) that corresponds to Class II or a higher class (or less than 50% of left ventricular ejection fraction (LVEF)) under New York Heart Association (NYHA) classification.
    * Uncontrolled hypertension (SBP/DBP >140/90 mmHg) (e.g., patient with SBP/DBP >140/90 mmHg despite the best care including optimizing the anti-hypertensive medication regimen)
    * History of hypertensive crisis or pre-existing hypertensive encephalopathy
    * Pulmonary hypertension
    * Myocardial infarction
    * Uncontrolled arrythmia
    * Unstable angina
14. Patients with any significant vascular diseases (e.g., aortic aneurysm requiring surgery or recent peripheral artery thrombosis) within 6 months prior to the initial treatment of the investigational product.
15. History of hypersensitivity reactions to any components of the investigational product or other drugs of the same class (humanized/human monoclonal antibody drugs)
16. Patients who are receiving any other investigational agents.
17. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab. Note: While enrolled, patients should not receive any live vaccines while receiving durvalumab and up to 30 days after last dose of durvalumab.
18. Patients who experience any grade 3-4 gastrointestinal (GI) bleeding within 3 months preceding Day 1
19. Diagnosis of hepatic encephalopathy
20. History of malignant bowel obstruction
21. Patients with psychiatric illness/social situations that would limit compliance with study requirements
22. Pregnant women are excluded from this study because CTX-009 is a recombinant bispecific antibody with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CTX-009, breastfeeding should be discontinued if the mother is treated with CTX-009. These potential risks may also apply to other agents used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ian Hu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org